CLINICAL TRIAL: NCT07158632
Title: Effects of Maternal Handwashing Education and Household Water Chlorination on Diarrheal Disease Among Under-Five Children in Central Ethiopia Using RCT
Brief Title: Effects of Multiple Interventions on Under-Five Diarrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Melaku Tesfaye, PhD Candidate, Jimma University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: JUIH/IRB/0509/25
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Diarrheal Diseases
Keywords: central Ethiopia, Diarrhea, Ethiopia, Multiple Interventions
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: The study contains four arms; these are handwashing education arm, water chlorination arm, combination arm, and control arm
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- handwashing education only arm (Experimental): Arm A: This arm receives handwashing education.
  Interventions: Behavioral: handwashing education
- water chlorination only arm (Experimental): Arm B: This arm receives household water chlorination
  Interventions: Behavioral: water chlorination
- combined hand washing and water chlorination arm (Experimental): Arm C: This arm receives both handwashing education and water chlorination.
  Interventions: Behavioral: combined intervention
- No intervention arm (No Intervention): This arm have not receive any intervention

INTERVENTIONS:
Behavioral: handwashing education — Arm A: This arm receive handwashing education using social and behavioral change communication
  Arms: handwashing education only arm
Behavioral: water chlorination — Arm B: This arm receives water chlorination intervention
  Arms: water chlorination only arm
Behavioral: combined intervention — Arm C: This arm receives combined handwashing and water chlorination intervention
  Arms: combined hand washing and water chlorination arm

SUMMARY:
Diarrhea is the leading cause of death, especially in developed nations. Though there are effective interventions, diarrhea remains the leading cause of death among children in Ethiopia

DETAILED DESCRIPTION:
Diarrheal disease is the major cause of child morbidity and mortality in low-income countries, including Ethiopia. Diarrhea is more common in areas with a lack of water sanitation and hygiene. Even though there are available effective interventions, diarrhea remains the major cause of child morbidity and mortality in Ethiopia. Therefore, the aim of this study is to give up-to-date information on multiple interventions that reduce diarrheal disease.

ELIGIBILITY:
Inclusion Criteria

* a child age from 6 to 59 months Exclusion Criteria
* severely ill mother, households that receive treated water

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 840 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of diarrhea among under-five children | At baseline and to four-month follow-up

SECONDARY OUTCOMES:
Adherence of interventions | Up to four-month follow-up
  percentage of soap availability near toilet and residual chlorine in drinking water

CONTACTS AND LOCATIONS:
Locations (1):
- Butajira Health Center, Butajīra, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breastfeeding and protection against diarrhea: an integrative review of literature Aleitamento materno e proteção contra diarreia: revisão integrativa da literatura Floriacy Stabnow Santos1 , Felipe César Stabnow Santos2 Adriana Moraes Leite1 , Leonardo Hunaldo dos Santos3 , Débora Falleiros de Mello1